CLINICAL TRIAL: NCT04193410
Title: Healthy Childcare Centre of the Future
Acronym: HCCF
Status: Completed | Type: Observational
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: METCZ20190144
Record Dates: First submitted 2019-12-03; First posted 2019-12-10 (Actual); Results first posted 2025-12-16 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2023-06

CONDITIONS: Health and Wellbeing of Primary School-aged Children
Keywords: Nutrition; Physical activity; School; Children; Prevention; School Health
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: Various health-promoting initiatives — No intervention is allocated in this study other than activities planned by childcare centres in accordance with wishes and needs of childcare centre staff and parents.

SUMMARY:
Rationale: In 2015-2020, the Dutch 'Healthy Primary School of the Future' intervention took place. Two schools became 'Healthy Primary Schools of the Future'; providing a healthy lunch and structured physical activity (PA) sessions. Two other 'Physical Activity Schools' only implemented the PA sessions. The intervention showed promising effects on children's BMI z-score and dietary and PA behaviours. Following these promising results, childcare centres of educational board Prisma have expressed their interest in implementing changes fitting the 'Healthy Primary School of the Future'. However, this is more complex than it seems to be, as budget to implement changes is lower and all childcare centres have a unique context. Therefore, there is a need to investigate how 'Healthy Primary School of the Future' can successfully be implemented in various, real-life school-settings. It is hypothesised that to maximise implementation and sustainability, each childcare centre will need to put together a set of changes and interventions which fit the context and needs of all stakeholders involved. No intervention is allocated in this study other than activities planned by childcare centres in accordance with wishes and needs of stakeholders.

Objective: To study the implementation of 'Healthy Childcare Centre of the Future' in different school-contexts and develop guidelines that can be used to facilitate widespread dissemination of the initiative. Secondary objectives include evaluating the initiative's effects on children's BMI z-score, general health, dietary and PA behaviours and school well-being. To reach these objectives, a process evaluation, effect evaluation and cost-effectiveness evaluation will be executed. Data will be collected using questionnaires (parents, children, teachers, directors), anthropometric measures (children), interviews (teachers, directors), observations and analyses of minutes of meetings.

DETAILED DESCRIPTION:
Rationale: From 2015-2020, the 'Healthy Primary School of the Future' intervention took place in Limburg, the Netherlands. The school environment of four primary schools changed. Two schools became 'Healthy Primary Schools of the Future'; providing their students with a healthy lunch and structured physical activity (PA) sessions during lunch time breaks. Two other 'Physical Activity Schools' only implemented the structured PA sessions. Interim analyses showed promising effects of the intervention; at two-year-follow-up, the study showed a significant decrease in BMI z-score of children in the 'Healthy Primary Schools of the Future' as compared with children in control schools. Also, positive intervention effects on dietary and PA behaviours were observed. Following these promising results, childcare centres of educational board Prisma have expressed their interest in implementing changes fitting the 'Healthy Primary School of the Future' initiative. However, this is more complex than it seems to be, as budget to implement changes is lower than in the original trial, and all childcare centres have a unique context. Therefore, there is a need to investigate how 'Healthy Primary School of the Future' can successfully be implemented in various, real-life school-settings. It is hypothesised that to maximise implementation and sustainability, each childcare centre will need to put together a set of changes and interventions which fit the context and needs of all stakeholders involved (e.g., the school board, teachers, parents and children).

Objective: The main objective is to study the implementation process of 'Healthy Childcare Centre of the Future' in different school-contexts and develop guidelines that can be used to facilitate widespread dissemination of the initiative. Secondary objectives include evaluating the effects of the 'Healthy Childcare Centre of the Future' on children's BMI z-score, general health, dietary and PA behaviours and school well-being. To reach these objectives, a process evaluation, effect evaluation and cost-effectiveness evaluation will be executed.

Study design: A non-randomised, non-controlled, observational study design. Study population: Children in study years four to six (at baseline) of twelve childcare centres located in Limburg, the Netherlands.

Main parameters/endpoints: The main study parameter of the effect evaluation is the change in absolute BMI z-score, which will be compared between the childcare centres categorised based on their degree of implementation (using categories based on the Diffusion of Innovations Theory).

Methods: Data will be collected in the form of questionnaires (parents, children, teachers/pedagogical employees, directors), anthropometric measurements (children), interviews (teachers/pedagogical employees, directors), observations and analyses of minutes of meetings.

Nature and extend of the burden and risks associated with participation: No intervention is allocated in this study other than activities planned by childcare centres in accordance with wishes and needs of childcare centre staff and parents. All outcome measures are non-invasive. The measurement protocol was designed while taking into account both a minimal burden for participants and a relevant scientific output for stakeholders (e.g., school board, teachers, parents/caregivers and children). Burden of participants is minimalised by incorporating most measurements in the regular school day.

ELIGIBILITY:
Inclusion Criteria:

* Student from study years four to six (at baseline) at one of the the predetermined childcare centres

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: A closed design will be used, meaning that at baseline (T0), all children in study year four to six of the childcare centres will be invited to participate in the study. At T1, these children will be students in study year five to seven, and at T2 they will be in study year six to eight. Based on the amount of children enrolled in school year 2019/2020, approximately 685 children are eligible to participate in the study.
Sampling Method: Non-Probability Sample
Enrollment: 315 (Actual)
Dates: Start 2020-06-15 (Actual); Primary Completion 2023-06-28 (Actual); Study Completion 2023-06-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marla Hahnraths, MSc, Principal Investigator — PhD candidate
Locations (1):
- Stichting Prisma, Panningen, Netherlands

IPD SHARING:
Plan to Share IPD: No
It is not our intention to share individual participant data with other researchers

REFERENCES:
- [Background] Bartelink NHM, Van Assema P, Jansen MWJ, Savelberg HHCM, Willeboordse M, Kremers SPJ. The Healthy Primary School of the Future: A Contextual Action-Oriented Research Approach. Int J Environ Res Public Health. 2018 Oct 12;15(10):2243. doi: 10.3390/ijerph15102243. PMID 30720796
- [Background] Willeboordse M, Jansen MW, van den Heijkant SN, Simons A, Winkens B, de Groot RH, Bartelink N, Kremers SP, van Assema P, Savelberg HH, de Neubourg E, Borghans L, Schils T, Coppens KM, Dietvorst R, Ten Hoopen R, Coomans F, Klosse S, Conjaerts MH, Oosterhoff M, Joore MA, Ferreira I, Muris P, Bosma H, Toppenberg HL, van Schayck CP. The Healthy Primary School of the Future: study protocol of a quasi-experimental study. BMC Public Health. 2016 Jul 26;16:639. doi: 10.1186/s12889-016-3301-9. PMID 27456845
- [Background] Bartelink NHM, van Assema P, Kremers SPJ, Savelberg HHCM, Oosterhoff M, Willeboordse M, van Schayck OCP, Winkens B, Jansen MWJ. Can the Healthy Primary School of the Future offer perspective in the ongoing obesity epidemic in young children? A Dutch quasi-experimental study. BMJ Open. 2019 Oct 31;9(10):e030676. doi: 10.1136/bmjopen-2019-030676. PMID 31676651
- [Background] Bartelink NHM, van Assema P, Kremers SPJ, Savelberg HHCM, Oosterhoff M, Willeboordse M, van Schayck OCP, Winkens B, Jansen MWJ. One- and Two-Year Effects of the Healthy Primary School of the Future on Children's Dietary and Physical Activity Behaviours: A Quasi-Experimental Study. Nutrients. 2019 Mar 22;11(3):689. doi: 10.3390/nu11030689. PMID 30909515

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: Schools
Groups:
- Medium implementers; Low implementers: As the present study investigated the effectiveness of health-promoting activities under real-world conditions and all participating schools were free to implement activities of their choice, there were no intervention or control groups. Instead, schools were categorised on the basis of the implemented activities' intensity. This resulted in the formation of two groups: medium implementers (six schools) and low implementers (five schools). The project's effectiveness on various health outcomes was compared between these two groups.
Period: Overall Study
Arm/Group | Medium implementers | Low implementers
Started | 143; 6 Schools | 172; 5 Schools
Completed | 136; 6 Schools | 166; 5 Schools
Not Completed | 7; 0 Schools | 6; 0 Schools
Not completed — Lost to Follow-up | 7 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Medium Implementers | Low Implementers | Total
Number analyzed (Participants) | 143 | 172 | 315
Age, Continuous [Mean (Standard Deviation); unit: years] | 9.21 (1.00) | 9.17 (0.96) | 9.19 (0.98)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 72 | 105 | 177
  Male | 71 | 67 | 138
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Population: The number analysed in this row differs from the overall number of participants, as we could not collect baseline data in all participants for this variable.
  Participants
    Western/Non-Western: number analyzed (Participants) | 131 | 152 | 283
    Western/Non-Western: Western | 125 | 149 | 274
    Western/Non-Western: Non-Western | 6 | 3 | 9
Study year [Count of Participants; unit: Participants]
  Four | 48 | 52 | 100
  Five | 37 | 62 | 99
  Six | 58 | 58 | 116
Socioeconomic status [Count of Participants; unit: Participants] — Population: The number analysed in this row differs from the overall number of participants, as we could not collect baseline data in all participants for this variable.
  Participants
    number analyzed (Participants) | 131 | 153 | 284
    Lowest tertile | 32 | 22 | 54
    Middle tertile | 39 | 47 | 86
    Highest tertile | 60 | 84 | 144
BMI z-score [Mean (Standard Deviation); unit: Z-score] — Children's Body Mass Index (BMI) was assessed by height and weight; age- and sex-specific BMI cut-off points were used to define overweight and obesity. BMI z-scores were calculated using Dutch reference values. A z-score of 0 represents the population mean. A z-score > 0 means a BMI higher than the population mean, a z-score of < 0 means a BMI lower than the population mean, both can pose specific health-related risks.
  Z-score | -0.15 (0.82) | -0.10 (0.94) | -0.13 (0.89)
Overweight/obese [Count of Participants; unit: Participants] — Children's Body mass index (BMI) was assessed by height and weight; age- and sex-specific BMI cut-off points were used to define overweight and obesity.
  Participants
    Overweight/obese | 43 | 21 | 64
    Normal weight | 100 | 151 | 251
Waist circumference [Mean (Standard Deviation); unit: centimeters] | 56.84 (4.66) | 58.62 (6.77) | 57.81 (5.96)
Physical activity summary score [Mean (Standard Deviation); unit: units on a scale] — The child questionnaire was used to gain insight into children's PA behaviour. The questionnaire contained ten items derived from the International Physical Activity Questionnaire for Children (IPAQ-C), which has acceptable validity. Activity scores between 1 and 5 were obtained for each item, after which the mean of these scores was calculated to obtain the total activity summary score (ranging from 1 (low PA) to 5 (high PA)).
  units on a scale | 3.04 (0.64) | 2.94 (0.67) | 2.98 (0.66)
Healthy dietary behaviours [Mean (Standard Deviation); unit: mean days/week] — A composite score for healthy dietary behaviours was computed from four separate questions. This score was calculated by averaging the weekly consumption (ranging from never (0) to every day (7)) of breakfast consumption and intake of fruit, warm and raw vegetables, and water throughout the day, as reported in the parental questionnaire.
  mean days/week | 5.57 (0.96) | 5.56 (0.95) | 5.56 (0.95)
Soft drink consumption [Mean (Standard Deviation); unit: mean days/week] — Soft drink consumption during the past week was derived from the parental questionnaire ranging from never (0) to every day (7).
  mean days/week | 4.31 (2.74) | 4.06 (2.78) | 4.17 (2.76)
School water consumption [Mean (Standard Deviation); unit: units on a scale] — Water consumption during school hours was derived from the child questionnaire ranging from never (0) to every day (3).
  units on a scale | 1.43 (1.22) | 1.25 (1.13) | 1.33 (1.17)
Fruit at lunch [Count of Participants; unit: Participants] — The child lunch questionnaire assessed children's consumption of certain food types during lunch. The items were summarised into six dichotomous (yes/no) food types: fruits, vegetables, grains (bread and cereals), dairy (milk/yoghurt and cheese), water, and butter.
  Participants
    %yes | 49 | 59 | 108
    %no | 94 | 113 | 207
Vegetables at lunch [Count of Participants; unit: Participants] — The child lunch questionnaire assessed children's consumption of certain food types during lunch. The items were summarised into six dichotomous (yes/no) food types: fruits, vegetables, grains (bread and cereals), dairy (milk/yoghurt and cheese), water, and butter.
  Participants
    %yes | 35 | 44 | 79
    %no | 108 | 128 | 236
Grains at lunch [Count of Participants; unit: Participants] — The child lunch questionnaire assessed children's consumption of certain food types during lunch. The items were summarised into six dichotomous (yes/no) food types: fruits, vegetables, grains (bread and cereals), dairy (milk/yoghurt and cheese), water, and butter.
  Participants
    %yes | 132 | 161 | 293
    %no | 11 | 11 | 22
Dairy at lunch [Count of Participants; unit: Participants] — The child lunch questionnaire assessed children's consumption of certain food types during lunch. The items were summarised into six dichotomous (yes/no) food types: fruits, vegetables, grains (bread and cereals), dairy (milk/yoghurt and cheese), water, and butter.
  Participants
    %yes | 53 | 58 | 111
    %no | 90 | 114 | 204
Water at lunch [Count of Participants; unit: Participants] — The child lunch questionnaire assessed children's consumption of certain food types during lunch. The items were summarised into six dichotomous (yes/no) food types: fruits, vegetables, grains (bread and cereals), dairy (milk/yoghurt and cheese), water, and butter.
  Participants
    %yes | 47 | 46 | 93
    %no | 96 | 126 | 222
Butter at lunch [Count of Participants; unit: Participants] — The child lunch questionnaire assessed children's consumption of certain food types during lunch. The items were summarised into six dichotomous (yes/no) food types: fruits, vegetables, grains (bread and cereals), dairy (milk/yoghurt and cheese), water, and butter.
  Participants
    %yes | 85 | 107 | 192
    %no | 58 | 65 | 123
At least two healthy food groups at lunch [Count of Participants; unit: Participants] — The child lunch questionnaire assessed children's consumption of certain food types during lunch. The items were summarised into six dichotomous (yes/no) food types: fruits, vegetables, grains (bread and cereals), dairy (milk/yoghurt and cheese), water, and butter. To shed more light on the nutritional value of the children's lunches, the different food types consumed were summed, and a dichotomous variable was created indicating whether children consumed at least two of the food types during lunch.
  Participants
    %yes | 125 | 152 | 277
    %no | 18 | 20 | 38

OUTCOME MEASURES:

1. Primary Outcome: BMI Z-score
Description: Children's Body Mass Index (BMI) was assessed by height and weight; age- and sex-specific BMI cut-off points were used to define overweight and obesity. BMI z-scores were calculated using Dutch reference values. A z-score of 0 represents the population mean. A z-score > 0 means a BMI higher than the population mean, a z-score of < 0 means a BMI lower than the population mean, both can pose specific health-related risks.
Time Frame: Two years
Population: The number analysed at T1 and T2 corresponds to the number of participants that were not LOF at T1 and T2.
Measure: Mean (Standard Deviation); unit: Z-score
Groups:
- Medium implementers: Participants from schools defined as medium implementers
- Low implementers: Participants defined as low implementers
Arm/Group | Medium implementers | Low implementers
Number analyzed (Participants) | 143 | 172
Z-score
  T0 (baseline) | -0.15 (0.82) | -0.10 (0.94)
  T1 (after one year): number analyzed (Participants) | 137 | 168
  T1 (after one year) | -0.14 (0.83) | -0.03 (0.97)
  T2 (after two years): number analyzed (Participants) | 136 | 166
  T2 (after two years) | -0.10 (0.88) | -0.05 (0.98)
Statistical Analysis 1: Comparison: Medium implementers vs Low implementers; Test type: Other — Linear mixed model analyses assessed longitudinal intervention effects on children's BMI z-score. A two-level model with measurements as first level and participants as second was used. The model's fixed part consisted of group (medium/low implementers), time (T0/T1/T2), interaction term of group with time, and covariates sex (boy/girl), study year at T0 (four/five/six), SES (low/middle/high), and children's weight status at T0 (underweight/normal weight/overweight). This analyses reports T1-T0; p = 0.210, Mixed Models Analysis
Statistical Analysis 2: Comparison: Medium implementers vs Low implementers; Linear mixed model analyses assessed longitudinal intervention effects on children's BMI z-score. A two-level model with measurements as first level and participants as second was used. The model's fixed part consisted of group (medium/low implementers), time (T0/T1/T2), interaction term of group with time, and covariates sex (boy/girl), study year at T0 (four/five/six), SES (low/middle/high), and children's weight status at T0 (underweight/normal weight/overweight). This analyses reports T2-T0; Test type: Other; p = 0.793, Mixed Models Analysis

2. Secondary Outcome: Mean Number of Days Per Week of Healthy Dietary Behaviours
Description: A composite score for healthy dietary behaviours was computed from four separate questions. This score was calculated by averaging the weekly consumption (ranging from never (0) to every day (7)) of breakfast consumption and intake of fruit, warm and raw vegetables, and water throughout the day, as reported in the parental questionnaire.
Time Frame: Two years
Population: The number analysed at T1 and T2 corresponds to the number of participants that were not LOF at T1 and T2.
Measure: Mean (Standard Deviation); unit: mean days/week
Arm/Group | Medium implementers | Low implementers
Number analyzed (Participants) | 114 | 142
mean days/week
  T0 (baseline) | 5.57 (0.96) | 5.56 (0.95)
  T1 (after one year): number analyzed (Participants) | 90 | 121
  T1 (after one year) | 5.38 (0.94) | 5.56 (0.90)
  T2 (after two years): number analyzed (Participants) | 82 | 119
  T2 (after two years) | 5.45 (0.90) | 5.52 (0.84)
Statistical Analysis 1: Comparison: Medium implementers vs Low implementers; Linear mixed model analyses were used to assess longitudinal intervention effects on children's dietary behaviours. A two-level model with measurements as first level and participants as second level was used. The model's fixed part consisted of group (medium/low implementers), time (T0/T1/T2), interaction term of group with time, and covariates sex (boy/girl), study year at baseline (four/five/six), SES (low/middle/high), and children's BMI z-score at baseline. This analysis reports T1-T0; Test type: Other; p = 0.444, Mixed Models Analysis
Statistical Analysis 2: Comparison: Medium implementers vs Low implementers; Linear mixed model analyses were used to assess longitudinal intervention effects on children's dietary behaviours. A two-level model with measurements as first level and participants as second level was used. The model's fixed part consisted of group (medium/low implementers), time (T0/T1/T2), interaction term of group with time, and covariates sex (boy/girl), study year at baseline (four/five/six), SES (low/middle/high), and children's BMI z-score at baseline. This analysis reports T2-T0; Test type: Other; p = 0.863, Mixed Models Analysis

3. Secondary Outcome: Child Physical Activity Behaviour (Child-reported)
Description: Assessed using the validated Physical Activity Questionnaire for Children (PAQ-C).The PAQ-C is a self-administered,7-day recall instrument, which provides a summary physical activity score derived from eight items, each scored on a 5-point scale. Item 1 (spare time activity) from no activity = 1; 7 times or more = 5. Items 2 to 7 (PE, lunch, right after school, evening, weekends) from lowest activity response = 1 or highest activity response = 5. Item 8 (mean of all days of the week) from none = 1; very often = 5. Item 9 (identifies students who are unusual active during the previous week). By adding up all means of the first eight items in PAQ-C, a summative score of physical activity is obtained. A score of 1 indicates low physical activity level, whereas a score of 5 indicates high physical activity level.
Time Frame: Two years
Population: The number analysed at T1 and T2 corresponds to the number of participants that were not LOF at T1 and T2.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Low implementers: Participants from schools defined as low implementers
Arm/Group | Medium implementers | Low implementers
Number analyzed (Participants) | 143 | 172
score on a scale
  T0 (baseline) | 3.04 (0.64) | 2.94 (0.67)
  T1 (after one year): number analyzed (Participants) | 137 | 168
  T1 (after one year) | 3.19 (0.58) | 3.25 (0.59)
  T2 (after two years): number analyzed (Participants) | 136 | 166
  T2 (after two years) | 3.12 (0.62) | 3.17 (0.65)
Statistical Analysis 1: Comparison: Medium implementers vs Low implementers; Linear mixed model analyses were used to assess longitudinal intervention effects on children's PA score. A two-level model with measurements as first level and participants as second level was used. The model's fixed part consisted of group (medium/low implementers), time (T0/T1/T2), interaction term of group with time, and covariates sex (boy/girl), study year at baseline (four/five/six), SES (low/middle/high), and children's BMI z-score at baseline. This analysis reports T1-T0; Test type: Other; p = 0.053, Mixed Models Analysis
Statistical Analysis 2: Comparison: Medium implementers vs Low implementers; Linear mixed model analyses were used to assess longitudinal intervention effects on children's PA score. A two-level model with measurements as first level and participants as second level was used. The model's fixed part consisted of group (medium/low implementers), time (T0/T1/T2), interaction term of group with time, and covariates sex (boy/girl), study year at baseline (four/five/six), SES (low/middle/high), and children's BMI z-score at baseline. This analysis reports T2-T0; Test type: Other; p = 0.209, Mixed Models Analysis

4. Secondary Outcome: Child Waist Circumference
Description: Waist circumference is measured with a measuring tape to the nearest 0.1 cm, following the World Health Organisation's assessment protocol.
Time Frame: Two years
Population: Number analysed at T1 and T2 corresponds to number of participants that were not LOF at T1 and T2.
Measure: Mean (Standard Deviation); unit: centimeters
Arm/Group | Medium implementers | Low implementers
Number analyzed (Participants) | 143 | 172
centimeters
  T0 (baseline) | 56.84 (4.66) | 58.62 (6.77)
  T1 (after one year): number analyzed (Participants) | 137 | 168
  T1 (after one year) | 58.49 (5.64) | 59.40 (6.68)
  T2 (after two years): number analyzed (Participants) | 136 | 166
  T2 (after two years) | 61.12 (5.94) | 61.57 (7.11)
Statistical Analysis 1: Comparison: Medium implementers vs Low implementers; Linear mixed model analyses were used to assess longitudinal intervention effects on children's waist circumference. A two-level model with measurements as first level and participants as second level was used. The model's fixed part consisted of group (medium/low implementers), time (T0/T1/T2), interaction term of group with time, and covariates sex (boy/girl), study year at baseline (four/five/six), SES (low/middle/high), and children's BMI z-score at baseline. This analysis reports T1-T0; Test type: Other; p = 0.003, Mixed Models Analysis
Statistical Analysis 2: Comparison: Medium implementers vs Low implementers; Linear mixed model analyses were used to assess longitudinal intervention effects on children's waist circumference. A two-level model with measurements as first level and participants as second level was used. The model's fixed part consisted of group (medium/low implementers), time (T0/T1/T2), interaction term of group with time, and covariates sex (boy/girl), study year at baseline (four/five/six), SES (low/middle/high), and children's BMI z-score at baseline. This analysis reports T2-T0; Test type: Other; p < 0.001, Mixed Models Analysis

5. Secondary Outcome: Mean Number of Days Per Week of Soft Drink Consumption
Description: Soft drink consumption during the past week was derived from the parental questionnaire ranging from never (0) to every day (7).
Time Frame: Two years
Population: The number analysed at T1 and T2 corresponds to the number of participants that were not LOF at T1 and T2.
Measure: Mean (Standard Deviation); unit: mean days/week
Arm/Group | Medium implementers | Low implementers
Number analyzed (Participants) | 114 | 142
mean days/week
  T0 (baseline) | 4.31 (2.74) | 4.06 (2.78)
  T1 (after one year): number analyzed (Participants) | 90 | 121
  T1 (after one year) | 4.07 (2.67) | 3.63 (2.88)
  T2 (after two years): number analyzed (Participants) | 82 | 119
  T2 (after two years) | 3.35 (2.61) | 3.43 (2.70)
Statistical Analysis 1: Comparison: Medium implementers vs Low implementers; [analysis description as in outcome 2, analysis 1]; Test type: Other; p = 0.815, Mixed Models Analysis
Statistical Analysis 2: Comparison: Medium implementers vs Low implementers; [analysis description as in outcome 2, analysis 2]; Test type: Other; p = 0.418, Mixed Models Analysis

6. Secondary Outcome: Water Consumption During School Hours
Description: Water consumption during school hours was derived from the child questionnaire ranging from never (0) to every day (3).
Time Frame: Two years
Population: The number analysed at T1 and T2 corresponds to the number of participants that were not LOF at T1 and T2.
Measure: Mean (Standard Deviation); unit: mean days/week
Arm/Group | Medium implementers | Low implementers
Number analyzed (Participants) | 143 | 172
mean days/week
  T0 (baseline) | 1.43 (1.22) | 1.25 (1.13)
  T1 (after one year): number analyzed (Participants) | 137 | 168
  T1 (after one year) | 1.47 (1.13) | 1.40 (1.16)
  T2 (after two years): number analyzed (Participants) | 136 | 166
  T2 (after two years) | 1.63 (1.20) | 1.73 (1.17)
Statistical Analysis 1: Comparison: Medium implementers vs Low implementers; [analysis description as in outcome 2, analysis 1]; Test type: Other; p = 0.307, Mixed Models Analysis
Statistical Analysis 2: Comparison: Medium implementers vs Low implementers; [analysis description as in outcome 2, analysis 2]; Test type: Other; p = 0.263, Mixed Models Analysis

7. Secondary Outcome: Fruit Consumption at Lunch
Description: The child lunch questionnaire assessed children's consumption of certain food types during lunch. The items were summarised into six dichotomous (yes/no) food types: fruits, vegetables, grains (bread and cereals), dairy (milk/yoghurt and cheese), water, and butter.
Time Frame: Two years
Population: The number analysed at T1 and T2 corresponds to the number of participants that were not LOF at T1 and T2.
Measure: Number; unit: percentage of yes
Arm/Group | Medium implementers | Low implementers
Number analyzed (Participants) | 143 | 172
percentage of yes
  T0 (baseline) | 34.3 | 34.3
  T1 (after one year): number analyzed (Participants) | 137 | 168
  T1 (after one year) | 31.4 | 26.8
  T2 (after two years): number analyzed (Participants) | 136 | 166
  T2 (after two years) | 22.8 | 23.5
Statistical Analysis 1: Comparison: Medium implementers vs Low implementers; Logistic mixed model analyses were used to assess longitudinal intervention effects on children's binary dietary behaviours. A two-level model with measurements as first level and participants as second level was used. The model's fixed part consisted of group (medium/low implementers), time (T0/T1/T2), interaction term of group with time, and covariates sex (boy/girl), study year at baseline (four/five/six), SES (low/middle/high), and children's BMI z-score at baseline. Analysis reports T1-T0; Test type: Other; p = 0.249, Mixed Models Analysis
Statistical Analysis 2: Comparison: Medium implementers vs Low implementers; Logistic mixed model analyses were used to assess longitudinal intervention effects on children's binary dietary behaviours. A two-level model with measurements as first level and participants as second level was used. The model's fixed part consisted of group (medium/low implementers), time (T0/T1/T2), interaction term of group with time, and covariates sex (boy/girl), study year at baseline (four/five/six), SES (low/middle/high), and children's BMI z-score at baseline. Analysis reports T2-T0; Test type: Other; p = 0.803, Mixed Models Analysis

8. Secondary Outcome: Vegetable Consumption at Lunch
Description: as for outcome 7
Time Frame: Two years
Population: The number analysed at T1 and T2 corresponds to the number of participants that were not LOF at T1 and T2.
Measure: Number; unit: percentage of yes
Arm/Group | Medium implementers | Low implementers
Number analyzed (Participants) | 143 | 172
percentage of yes
  T0 (baseline) | 24.5 | 25.6
  T1 (after one year): number analyzed (Participants) | 137 | 168
  T1 (after one year) | 31.4 | 26.8
  T2 (after two years): number analyzed (Participants) | 136 | 166
  T2 (after two years) | 19.9 | 19.9
Statistical Analysis 1: Comparison: Medium implementers vs Low implementers; [analysis description as in outcome 7, analysis 1]; Test type: Other; p = 0.073, Mixed Models Analysis
Statistical Analysis 2: Comparison: Medium implementers vs Low implementers; [analysis description as in outcome 7, analysis 2]; Test type: Other; p = 0.658, Mixed Models Analysis

9. Secondary Outcome: Grain Consumption at Lunch
Description: as for outcome 7
Time Frame: Two years
Population: The number analysed at T1 and T2 corresponds to the number of participants that were not LOF at T1 and T2.
Measure: Number; unit: percentage of yes
Arm/Group | Medium implementers | Low implementers
Number analyzed (Participants) | 143 | 172
percentage of yes
  T0 (baseline) | 92.3 | 93.6
  T1 (after one year): number analyzed (Participants) | 137 | 168
  T1 (after one year) | 94.2 | 93.5
  T2 (after two years): number analyzed (Participants) | 136 | 166
  T2 (after two years) | 94.9 | 92.8
Statistical Analysis 1: Comparison: Medium implementers vs Low implementers; [analysis description as in outcome 7, analysis 1]; Test type: Other; p = 0.742, Mixed Models Analysis
Statistical Analysis 2: Comparison: Medium implementers vs Low implementers; [analysis description as in outcome 7, analysis 2]; Test type: Other; p = 0.370, Mixed Models Analysis

10. Secondary Outcome: Dairy Consumption at Lunch
Description: as for outcome 7
Time Frame: Two years
Population: The number analysed at T1 and T2 corresponds to the number of participants that were not LOF at T1 and T2.
Measure: Number; unit: percentage of yes
Arm/Group | Medium implementers | Low implementers
Number analyzed (Participants) | 143 | 172
percentage of yes
  T0 (baseline) | 37.1 | 33.7
  T1 (after one year): number analyzed (Participants) | 137 | 168
  T1 (after one year) | 39.4 | 39.3
  T2 (after two years): number analyzed (Participants) | 136 | 166
  T2 (after two years) | 48.5 | 38.0
Statistical Analysis 1: Comparison: Medium implementers vs Low implementers; [analysis description as in outcome 7, analysis 1]; Test type: Other; p = 0.483, Mixed Models Analysis
Statistical Analysis 2: Comparison: Medium implementers vs Low implementers; [analysis description as in outcome 7, analysis 2]; Test type: Other; p = 0.626, Mixed Models Analysis

11. Secondary Outcome: Water Consumption at Lunch
Description: as for outcome 7
Time Frame: Two years
Population: The number analysed at T1 and T2 corresponds to the number of participants that were not LOF at T1 and T2.
Measure: Number; unit: percentage of yes
Arm/Group | Medium implementers | Low implementers
Number analyzed (Participants) | 143 | 172
percentage of yes
  T0 (baseline) | 32.9 | 26.7
  T1 (after one year): number analyzed (Participants) | 137 | 168
  T1 (after one year) | 38.0 | 31.0
  T2 (after two years): number analyzed (Participants) | 136 | 166
  T2 (after two years) | 44.9 | 38.6
Statistical Analysis 1: Comparison: Medium implementers vs Low implementers; [analysis description as in outcome 7, analysis 1]; Test type: Other; p = 0.771, Mixed Models Analysis
Statistical Analysis 2: Comparison: Medium implementers vs Low implementers; [analysis description as in outcome 7, analysis 1]; Test type: Other; p = 0.861, Mixed Models Analysis

12. Secondary Outcome: Butter Consumption at Lunch
Description: as for outcome 7
Time Frame: Two years
Population: The number analysed at T1 and T2 corresponds to the number of participants that were not LOF at T1 and T2.
Measure: Number; unit: percentage of yes
Arm/Group | Medium implementers | Low implementers
Number analyzed (Participants) | 143 | 172
percentage of yes
  T0 (baseline) | 59.4 | 62.2
  T1 (after one year): number analyzed (Participants) | 137 | 168
  T1 (after one year) | 59.1 | 60.7
  T2 (after two years): number analyzed (Participants) | 136 | 166
  T2 (after two years) | 55.1 | 56.6
Statistical Analysis 1: Comparison: Medium implementers vs Low implementers; [analysis description as in outcome 7, analysis 1]; Test type: Other; p = 0.766, Mixed Models Analysis
Statistical Analysis 2: Comparison: Medium implementers vs Low implementers; [analysis description as in outcome 7, analysis 2]; Test type: Other; p = 0.995, Mixed Models Analysis

13. Secondary Outcome: Consumption of at Least Two Healthy Food Groups During Lunch
Description: The child lunch questionnaire assessed children's consumption of certain food types during lunch. The items were summarised into six dichotomous (yes/no) food types: fruits, vegetables, grains (bread and cereals), dairy (milk/yoghurt and cheese), water, and butter. To shed more light on the nutritional value of the children's lunches, the different food types consumed were summed, and a dichotomous variable was created indicating whether children consumed at least two of the food types during lunch.
Time Frame: Two years
Population: The number analysed at T1 and T2 corresponds to the number of participants that were not LOF at T1 and T2.
Measure: Number; unit: percentage of yes
Arm/Group | Medium implementers | Low implementers
Number analyzed (Participants) | 143 | 172
percentage of yes
  T0 (baseline) | 87.4 | 88.4
  T1 (after one year): number analyzed (Participants) | 137 | 168
  T1 (after one year) | 86.1 | 88.7
  T2 (after two years): number analyzed (Participants) | 136 | 166
  T2 (after two years) | 89.7 | 86.7
Statistical Analysis 1: Comparison: Medium implementers vs Low implementers; [analysis description as in outcome 7, analysis 1]; Test type: Other; p = 0.437, Mixed Models Analysis
Statistical Analysis 2: Comparison: Medium implementers vs Low implementers; [analysis description as in outcome 7, analysis 1]; Test type: Other; p = 0.798, Mixed Models Analysis

ADVERSE EVENTS:
Time Frame: One year after baseline and two years after baseline.
Description: As there was no intervention administered as part of the study, there was no risk for all-cause mortality or (serious) adverse effects as part of the study.
Groups:
- All participants: As there were no intervention and control groups included in the present study, participants were not categorised in different arms/groups. This arm/group therefore includes all participants in the study.
Arm/Group | All participants
All-Cause Mortality (participants affected / at risk) | 0/315
Serious Adverse Events (participants affected / at risk) | 0/315
Other Adverse Events (participants affected / at risk) | 0/315

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-02-04): https://cdn.clinicaltrials.gov/large-docs/10/NCT04193410/Prot_SAP_000.pdf